CLINICAL TRIAL: NCT00901602
Title: Lebanese Interhospital Pneumococcal Surveillance Program (LIPSP)
Brief Title: Lebanese Interhospital Pneumococcal Surveillance Program
Acronym: LIPSP
Status: Recruiting | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: PneumoADIP (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Ghassan Dbaibo, Professor, American University of Beirut Medical Center
Other Study IDs: PNEUMOSurv1LIPSP
Record Dates: First submitted 2009-05-08; First posted 2009-05-14 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia; Meningitis; Sepsis; Bacteremia
Keywords: streptococcus pneumoniae; pneumococcus; pneumonia; meningitis; serotypes; bacteremia; sepsis
MeSH Terms: conditions — Pneumonia; Meningitis; Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
Streptococcus pneumoniae (pneumococcus) is a bacterium that causes severe infections in children and adults such as meningitis, pneumonia, and blood stream infection. There are many types of these bacteria defined by the type of sugar coat that they have. These are classified as serotypes. There are common serotypes that cause severe disease and are preventable by vaccination of children. Other less common types are more difficult to prevent. The investigators aim to determine the serotypes that cause invasive pneumococcal disease in Lebanon and to study their sensitivity to different antibiotics. The investigators will collect bacterial isolates from different hospitals in Lebanon isolated from the blood or spinal fluid of patients with invasive pneumococcal disease. This information will help the investigators determine the usefulness of available pneumococcal vaccines in preventing these infections. The data will be distributed to all primary care physicians treating children in Lebanon and will be shared with the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Samples included in the study are those that are:

  * culture proven
  * invasive pneumococcal infections
  * in patients of all ages admitted to different hospitals all over Lebanon
* Acceptable samples include:

  * positive isolates from blood
  * cerebrospinal fluid
  * other normally sterile body sites such as empyema fluid, abscesses, joint fluid, middle ear fluid obtained by tympanocentesis in the operating room, and lung needle aspiration

Exclusion Criteria:

* non S. pneumoniae isolates

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with invasive pneumococcal disease with positive culture of S. pneumoniae from a normally sterile site (blood, CSF, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2005-10; Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Serotype prevalence of S. pneumoniae in invasive pneumococcal disease | yearly

SECONDARY OUTCOMES:
Determine the antibiotic sensitivity of S. pneumoniae and the association with specific serotypes | yearly

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan S Dbaibo, M.D., Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon